CLINICAL TRIAL: NCT06542822
Title: Immediate Effects of Intravenous Iron Therapy in Patients With Systolic Heart Failure and Iron Deficiency as Evaluated by Cardiac Magnetic Resonance Imaging: An Observational Prospective Study
Brief Title: IRONHEART: Intravenous Iron in Non-ischaemic Heart Failure
Acronym: IRONHEART
Status: Recruiting | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: RHMCAR0640
Record Dates: First submitted 2024-07-02; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure; Iron Deficiencies
Keywords: Ferric derisomaltose; Non-ischaemic heart failure; Chronic heart failure; Iron deficiency; Left ventricular failure; Iron homeostasis; Cardiac MRI; Cardiac Magnetic resonance imaging
MeSH Terms: conditions — Heart Failure; Iron Deficiencies | interventions — ferric derisomaltose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- IRONHEART Observational Study Group: 16 participants, with non-ischaemic heart failure, with iron deficiency TSATS <20% and heart failure with a reduced ejection fraction <40%.
  Cohort will have to be established on guideline directed heart failure therapy. Participants meeting eligibility criteria will undergo baseline quality of life questionnaires, hand grip tests and six minute walk tests before receiving intravenous iron derisomaltose and repeating these investigations again after 24 hours and 30 days including a cardiac magnetic resonance imaging.
  Interventions: Drug: Ferric derisomaltose

INTERVENTIONS:
Drug: Ferric derisomaltose — See group descriptions

SUMMARY:
The aim of this study is to observe the effect of intravenous ferric derisomaltose in participants with non-ischaemic heart failure (LVEF<40%), iron deficiency (TSATS<20%) and established on heart failure therapy including Sodium-glucose cotransporter 2 inhibitors (SGLT2i). Participants will undergo baseline laboratory blood tests, cardiac magnetic resonance imaging (cMRI), six-minute walk test, musculoskeletal function test and Kansas City Cardiomyopathy Questionnaire (KCCQ). These investigations will be repeated at 24 hours and 30 days after the administration of intravenous ferric derisomaltose.

DETAILED DESCRIPTION:
Heart failure is a neuro-endocrine syndrome in which patients report symptoms of breathlessness and lethargy accompanied with signs of fluid overload.

Iron deficiency is very common in heart failure, affecting up to 50% of patients. Its presence in this population is associated with worsening symptoms and increased risk of death. Human clinical trials have shown that administering intravenous iron improves quality of life and exercise tolerance. The European Society Guidelines gives a 1A class recommendation for intravenous iron replacement in symptomatic heart failure patients.

Iron is an essential micro-nutrient required in mitochondrial metabolism, handling of reactive oxygen species and cellular metabolism. Heart failure leads to a pro inflammatory state, resulting in reduced gastrointestinal absorption, and inhibition of iron mobilisation. Mouse models have shown reversal of cardiac fibrosis, cardiac remodelling, and reduction in the pro inflammatory state when treated with intravenous iron. Similarly iron deficient human cardiomyocytes show adverse remodelling and altered function reversed with iron repletion.

The investigators aim to recruit 16 participants with non-ischaemic heart failure, established on optimal medical therapy, including SGLT2i therapy, for four weeks prior to the start of the trial. Initial baseline investigations will include: cMRI, six-minute walk test, hand grip strength test, laboratory blood tests and a KCCQ-12. Intravenous ferric derisomaltose will be given as standard of care. These investigations will be repeated at 24 hours and at 30 days after the administration of intravenous ferric derisomaltose.

The study aims to observe changes pre and post administration of intravenous derisomaltose in the following:

* Changes in cardiac function and parametric measurements (T1/T2) as assessed by cardiac magnetic resonance imaging.
* Changes in high sensitivity troponin, N Terminal pro-Brain Natriuretic Peptide (NT pro-BNP) and serum phosphate levels.
* Changes in the submaximal exercise test (six-minute walk) and musculoskeletal function test (hand grip test).
* Changes in heart failure symptoms as assessed by KCCQ Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Participants capable of giving informed consent.
* Aged 18yrs and above.
* Diagnosed with heart failure and a reduction of their ejection fraction < 40% by any modality.
* Non ischaemic cardiomyopathy as determined by baseline cardiac magnetic resonance imaging.
* Iron deficient per this definition: Transferrin saturations < 20%.
* Established on Heart failure therapy including SGLT2i therapy for a minimum of four weeks prior to recruitment.
* New York Heart Association score of I - III class.

Exclusion Criteria:

* New York Heart Association classification Score >IV
* Ischaemic cardiomyopathy
* Chronic kidney stage: Estimated Glomerular Filtration Rate (eGFR) < 30
* Requirement for renal dialysis
* Atrial fibrillation / atrial flutter
* Non cardiac and cardiac palliative diagnosis
* Active cancer diagnosis
* Moderate to severe valvular heart disease
* Cardiac electronic implantable device: Cardiac resynchronization therapy, Implantable cardioverter-defibrillator, left ventricular assist device
* Cardiac & non cardiac transplant participants
* Myocardial infarction, Percutaneous Coronary Intervention, Coronary Artery Bypass Graft surgery in the last 30 days
* Complex congenital heart disease
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with non-ischaemic cardiomyopathy with a left ventricular function less than 40% and iron deficient as per the following criteria: Transferrin saturations < 20%
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Ejection Fraction quantified on Cardiac Magnetic Resonance Imaging | 24 Hours and 30 days
  Changes in Ejection Fraction quoted in (%)

SECONDARY OUTCOMES:
T1 Mapping quantified on Cardiac Magnetic Resonance Imaging | 24 Hours and 30 days
  Changes in T1 Parametric Mapping quantified in (msec)
T2 Mapping quantified on Cardiac Magnetic Resonance Imaging | 24 Hours and 30 Days
  Changes in T2 Parametric Mapping quantified in (msec)
Extracellular Volume (ECV) Fraction quantified on Cardiac Magnetic Resonance Imaging | 24 Hours and 30 Days
  Changes in ECV Fraction quoted in (%)
Ventricular Volumes quantified on Cardiac Magnetic Resonance Imaging | 24 Hours and 30 Days
  Changes in left and right ventricular volumes quantified in (ml)
Indexed Ventricular Volume quantified on Cardiac Magnetic Resonance Imaging | 24 Hours and 30 Days
  Changes in indexed left and right ventricular volumes. Weight and Height will be combined to calculate Body Surface Area (m2). Left Ventricular Volume in (ml) will be divided by Body Surface Area to give indexed value (ml/m2)
Strain analysis as quantified on Cardiac Magnetic Resonance Imaging | 24 Hours and 30 Days
  Changes in strain as assessed by feature tracking on cardiac magnetic resonance imaging
Quality of Life assessment: KCCQ-12 questionnaire | 24 Hours and 30 Days
  Changes in Kansas City Cardiomyopathy Questionnaire. Four sub-domains: Physical limitation, Symptom Frequency, Quality of life and social limitations. Scores range from 0 - 100, with higher scores reflecting a better heart status.
Submaximal Exercise Test: Six Minute Walk Test | 24 Hours and 30 Days
  Changes in distance walked (meters) in six minutes
Musculoskeletal function test: Hand grip test | 24 Hours and 30 Days
  Changes in Isometric Grip Force in (KG)
Haemoglobin | 30 Days
  Laboratory Blood Test
High Sensitivity troponin | 24 Hours and 30 Days
  Laboratory Blood Test
Phosphate | 24 Hours and 30 Days
  Laboratory Blood Test
N-terminal pro B type natriuretic peptide (NTproBNP) | 30 Days
  Laboratory Blood Test

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Flett, MBBS BSc MD, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire, United Kingdom